CLINICAL TRIAL: NCT03706014
Title: Innovative Family Prevention With Latino Siblings in Disadvantaged Settings
Acronym: SIBS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard University (Other)
Responsible Party: Principal Investigator, Adriana Umaña-Taylor, Professor, Harvard University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SITE18-0185
Record Dates: First submitted 2018-08-26; First posted 2018-10-15 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Promotion of Positive Sibling Relationships
Keywords: siblings; family; Latinos; social emotional competencies; parenting; middle childhood; late childhood

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial involving a contact-equivalent control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SIBS Program (Experimental): The program condition includes 12 weekly 90-minute afterschool group sessions for siblings. Sessions are structured as psycho-educational groups and include social interactional activities, role-playing, discussion, and didactic presentation. The focus is on sibling relationship skills, cognitions, and activities. During a total of 3 family nights, parents attend with their children. Part of the family night session involves parents and children together. Another part of the session involves parents being separated from children. Family Nights promote parents' understanding of sibling relationships, review concepts, provide strategies for parental support of siblings, and teach parents skills for dealing with sibling problems. Family Nights include dinner and last 2 hours.
  Interventions: Behavioral: SIBS Program
- Contact-Equivalent Attention Control (Placebo Comparator): The Contact-Equivalent Attention Control condition includes 12 weekly 90-minute afterschool group sessions for siblings led by two co-leaders. Students work on educational games and activities. Groups begin with an icebreaker and continue with games and projects. This condition also includes 3 family nights, where parents attend with their children. Activities of the Family Nights include children showing their parents the activities they have been engaging in during the sessions. Family Nights include dinner and last 2 hours. Part of the family night session involves parents and children together. Another part of the session involves parents being separated from children; during this part, parents will break out with one group leader, and siblings will work with the other group leader.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: SIBS Program — Universal prevention program promoting positive sibling and family relationships conducted in an afterschool setting
  Arms: SIBS Program
Behavioral: Control — Contact-equivalent attention control program in which students play educational games
  Arms: Contact-Equivalent Attention Control

SUMMARY:
The current study is a randomized intervention trial that tests the efficacy of a family-focused sibling relationship promotion program. The study includes a treatment group and a contact-equivalent attention control condition with 288 sibling dyads and data collection with target parents, target sibling dyads, and teachers at three time points (pre-test, post-test, and 18-month follow-up). Data will be collected using a three-cohort design with 96 families in each of the three cohorts.

DETAILED DESCRIPTION:
The proposed project tests the efficacy of a family-focused program. This innovative program is focused on sibling relationships and parenting of siblings as synergistic targets of change to promote positive interpersonal family dynamics and parent and youth psychosocial and behavioral health and well-being. This translational effort builds on strong theoretical and empirical premises including a successful pilot study (ASU SIBS Program). Using a rigorous design and measurement, aims are to: (a) test the efficacy of SIBS, delivered via 12 weekly afterschool sibling sessions and 3 family nights in the familiar elementary school setting, versus a contact-equivalent attention control condition. Mexican-origin sibling dyads (5th graders and younger siblings; N = 288 dyads) and their parents will be recruited from economically disadvantaged elementary schools and randomly assigned within school to intervention or contact-equivalent attention control conditions. Assessments will be conducted at pre-test, post-test, and 18-month follow-up. Program effects will be tested on primary and secondary outcomes, including sibling relationship quality (i.e., warmth and negativity), sibling relationship skills, children's efficacy (social, emotional), children's internalizing symptoms, parents' stress and depressive symptoms, parent-child warmth and conflict, and family cohesion. Findings will advance prevention science by identifying an efficacious program that capitalizes on cultural assets to promote positive family dynamics and psychosocial well-being among Latinos, including by incorporating daily measurements of intervention targets (sibling relationship skills) to identify mechanisms underlying program effects.

ELIGIBILITY:
Inclusion Criteria:

* Target child has to be a 5th grader
* Target child has to be of Latino/Hispanic heritage
* Target child has to have a younger sibling enrolled in the same school in the 1st through 4th grade
* Target child and younger sibling have to be enrolled students in a participating elementary school.

Exclusion Criteria:

- Enrollment in a self-contained special education setting

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2018-09-29 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Parenting of Siblings Measure | 16 weeks
  The measure assesses parents' perceptions of three constructs: Parents' positive guidance, authoritarian control, and involvement (McHale et al., 2000; Updegraff et al., 2016). For each subscale, scores range from 1 to 5. Higher subscale scores indicate more positive guidance (i.e., better outcome), higher involvement (i.e., better outcome), and higher authoritarian control (i.e., worse outcome). Subscales are not combined into a total score.
Sibling Prosocial Behavior | 16 weeks
  The measure assesses parents' perceptions of one construct: Parents' ratings of children's supportive and prosocial behaviors (Stormshak, Bellanti, & Bierman, 1996; Updegraff et al., 2016).
  Scores range from 1 to 6. Higher scores indicate parents' perceptions of target child's more prosocial behaviors toward their sibling (i.e., better outcome).
Sibling Intimacy | 16 weeks
  The measure assesses siblings' ratings of intimacy/emotional support (Blyth & Foster-Clark, 1987). Scores range from 1 to 5. Higher scores indicate target child's perceptions of higher sibling intimacy and closeness (i.e., better outcome).
Sibling Relationship Inventory: Negativity Subscale | 16 weeks
  The measure assesses parents' ratings of sibling conflict and negativity (Stocker & McHale, 1992). Scores range from 1 to 5. Higher scores indicate parents' perceptions of target child's greater negativity toward their sibling (i.e., worse outcome).
Sibling Relationship Inventory: Negativity Subscale | 16 weeks
  The measure assesses children's ratings of sibling conflict and negativity (Furman & Buhrmester, 1985). Scores range from 1 to 5. Higher scores indicate target child's perceptions of higher sibling conflict and negativity (i.e., worse outcome).

SECONDARY OUTCOMES:
Self-efficacy Measure | 16 weeks
  This measure assesses children's ratings of two constructs: social self-efficacy and emotional self-efficacy (Muris, 2001). For each subscale, scores range from 1 to 5. Higher subscale scores indicate greater social self-efficacy (i.e., better outcome) and greater emotional self-efficacy (i.e., better outcome). Subscales are not combined into a total score.
Children's Depression Inventory | 16 weeks
  This measure assesses children's ratings of their depressive symptoms (Kovacs, 1985). Items are scored on a scale from 0 to 2, and higher scores indicate greater depressive symptoms (i.e., worse outcome). If mean scores are used, scores range from 0 to 2. If sum scores are used, scores range from 0 to 52.
Behavior Problem Index | 16 weeks
  This measure assesses parents' perceptions of children's social emotional functioning in 6 domains (i.e., antisocial, anxious/depressed, headstrong, hyperactive, dependency, peer conflict; Peterson & Zill, 1986). For all scales, items are scored on a scale from 1 to 3. For each subcale, higher scores indicate higher problem behavior in the domain (i.e., worse outcome). Mean scores are created for each subscale, and a total mean score is created across all domains - in all cases, higher scores indicate worse outcomes.
Center for Epidemiological Depression Scale | 16 weeks
  The CES-D (Radloff, 1977) assesses parents' depressive symptoms. Items are scored on a scale from 0 to 3, and higher scores indicate greater depressive symptoms (i.e., worse outcome). No subscales are created. If mean scores are used, scores range from 0 to 3. If sum scores are used, scores range from 0 to 60.
Parenting Stress Index | 16 weeks
  This measure assesses parents' perceptions of parental stress and includes two subscales: parental distress and dysfunctional interaction (Abidin, 1995). Items for each subscale are scored on a scale from 1 to 5. Mean scores can be created for each subscale, and higher scores indicate higher levels of distress (i.e., worse outcome) and higher dysfunctional interaction (i.e., worse outcome). A total scale score can be created across all items and higher scores indicate higher parenting stress (i.e., worse outcome).
Children's Reports of Parental Behavior Inventory - Parent-Child Warmth | 16 weeks
  This measure assesses parent and child's report of parent-child warmth (Schaefer, 1965). Items are scored on a scale of 1 to 5. Items are average and higher scores indicate greater perceptions of parent-child warmth (i.e., better outcome).
Children's Reports of Parental Behavior Inventory - Harsh Discipline | 16 weeks
  This measure assesses parent's reports of harsh discipline (Schaefer, 1965). Items are scored on a scale of 1 to 5. Items are average and higher scores indicate greater perceptions of harsh discipline (i.e., worse outcome).
Parent-Child Conflict measure | 16 weeks
  This measure assesses parents' perceptions of parent-child conflict (Smetana, 1988). Items are scored on a scale from 1 to 6. Average scores are created and higher values indicate greater parent-child conflict (i.e., worse outcome).
Family Adaptability and Cohesion Evaluation Scales II | 16 weeks
  This measure assesses parents' perceptions of family cohesion (Olson, Portner, & Bell, 1982). Items are scored on a scale from 1 to 5. An average score is created and higher scores indicate greater family cohesion (i.e., better outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Adriana J Umana-Taylor, PhD, Principal Investigator — Harvard University; Kimberly A Updegraff, PhD, Principal Investigator — Arizona State University
Locations (1):
- Arizona State University, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Updegraff KA, Umana-Taylor AJ, Rodriguez De Jesus SA, McHale SM, Feinberg MF, Kuo SI. Family-focused prevention with Latinos: What about sisters and brothers? J Fam Psychol. 2016 Aug;30(5):633-40. doi: 10.1037/fam0000200. Epub 2016 Apr 14. PMID 27077238
- [Background] Feinberg ME, Solmeyer AR, Hostetler ML, Sakuma KL, Jones D, McHale SM. Siblings are special: initial test of a new approach for preventing youth behavior problems. J Adolesc Health. 2013 Aug;53(2):166-73. doi: 10.1016/j.jadohealth.2012.10.004. Epub 2012 Nov 20. PMID 23298985

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2021-03-23): https://cdn.clinicaltrials.gov/large-docs/14/NCT03706014/Prot_ICF_002.pdf
  • Statistical Analysis Plan (2018-10-10): https://cdn.clinicaltrials.gov/large-docs/14/NCT03706014/SAP_000.pdf